CLINICAL TRIAL: NCT04303182
Title: Laparoendoscopic Single-site Versus Three Port Totally Extraperitoneal Hernia Repair: A Prospective Double Blinded Randomized Clinical Trial
Brief Title: LESS TEP vs. Three Port TEP for Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sofia Med Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204
Record Dates: First submitted 2020-02-26; First posted 2020-03-10 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Inguinal Hernia
Keywords: TEP; LESS TEP; Inguinal Hernia; Laparoscopic Surgery; Recurrence inguinal hernia; Primary inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard 3 port TEP (Active Comparator): Group A will undergo laparoscopic TEP inguinal hernia repair with 3 ports (10 mm , and 2 ports of 5 mm ).
  Interventions: Procedure: Standard 3 port TEP
- LESS TEP (Active Comparator): Group B will undergo laparoscopic TEP inguinal hernia repair with a single skin incision 2-3cm.
  Interventions: Procedure: LESS TEP

INTERVENTIONS:
Procedure: Standard 3 port TEP — 3 port TEP inguinal hernia repair with 10mm. port under the umbilicus and two 5mm. port in line under the 10mm. port
  Arms: Standard 3 port TEP
Procedure: LESS TEP — TEP inguinal hernia repair with one vertical skin incision under the umbilicus
  Arms: LESS TEP

SUMMARY:
This study aim to compare efficacy and safety of Laparoendoscopic single site total extraperitoneal inguinal hernia repair /LESS TEP/ and traditional total extraperitoneal hernia repair with 3 ports /TEP/.

DETAILED DESCRIPTION:
This is a prospective, double blinded, randomized trial. It compared of Laparoendoscopic single site total extraperitoneal inguinal hernia repair /LESS TEP/ and traditional total extraperitoneal hernia repair with 3 ports /TEP/.

Inguinal hernia is one of the most common surgical diseases. Laparoscopic hernia repairs include two types, TEP and TAPP. Laparoscopic inguinal hernia repair was associated with less post operative pain, a shorter recovery period and better cosmetic results. Efforts are continuing to further reduce the port related morbidities and improve the cosmetic outcomes of laparoscopic surgery, including reduction of the size and number of ports. This has led to the evolution of a novel surgical approach now collectively known as laparoendoscopic single-site surgery.

200 patients will undergo TEP inguinal hernia repair. They will be randomized in two groups by sealed envelope method.

Group A: Standard TEP with 3 ports (10mm. and 2 ports of 5mm.). In case of difficulty in Standard 3 port TEP inguinal hernia repair, the procedure will be converted to TAPP.

Group B: LESS TEP with single skin incision 2-3cm. In case of difficulty in LESS TEP inguinal hernia repair, the procedure will be converted to standard 3 port repair or TAPP.

Patient will be informed at consenting that 3 wound plasters will be applied to their abdomen regardless of whether they are in the single port or 3- ports group so that they would not know which group they have been randomized to. The blind will only be lifted after pain score and area of pain has been recorded before discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Willing to participate in this study and signed an informed consent.
* Diagnosed inguinal hernia - primary or recurrence
* ASA class I, II and III

Exclusion Criteria:

* Age under 18 years and above 90 years
* Strangulated hernia
* Patients with severe chronic diseases or cardiopulmonary dysfunction, who can't undergo general anesthesia
* Patients who prefer a certain surgical approach
* Patients who undergo surgery procedures for chronic pain after inguinal hernia repair

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 24hours
  Assessment of post-operative pain according to the visual analog scale pain score - From 0 to 10 - 0 is no pain and 10 is severe pain.
Postoperative Pain | 1 week
  Assessment of post-operative pain according to the visual analog scale pain score - From 0 to 10 - 0 is no pain and 10 is severe pain.

SECONDARY OUTCOMES:
Operating time | During operation
Intraoperative complications | During operation
  Assessment of interoperation procedure of the incident of spermaduct, vessel and other organ damage
Length of hospital stay | 24 hours
Postoperative complications | 1 week; 4 weeks
  Urinary infections; Seroma; Hematoma
Recurrence of hernia | 4 weeks; 3 months; 1 year
Cosmetic scar score | 4 weeks
  Scar evaluation using Patient and Observer Scar Assessment Scale (POSAS) 4 week after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sofiamed Hospital, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No